CLINICAL TRIAL: NCT03756779
Title: Randomized, Cross-over Pilot Study of Blood Cholesterol Response to Dietary Saturated Fat in Patients With Autosomal Dominant Hypercholesterolemia
Brief Title: Cross-over Pilot Study of Blood Cholesterol Response to Dietary Saturated Fat in Patients With Autosomal Dominant Hypercholesterolemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enrolling subjects in the study.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 122016-032
Record Dates: First submitted 2017-07-28; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Familial Hypercholesterolemia
Keywords: Diet study
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Saturated Fat Diet (Experimental): Goal will be to attain <7% of daily calories from saturated fat. Replace it with energy from monounsaturated fat.
  Interventions: Other: Dietary intervention
- High Saturated Fat Diet (Active Comparator): Goal will be to attain 15% of daily calories from saturated fat. Decrease intake of monounsaturated fat.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Dietary intervention with dietary modification of fat intake.

SUMMARY:
We are performing a pilot cross-over diet study involving 5 patients with heterozygous FH and 5 patients with unexplained ADH. The patients will be randomized to a low versus high saturated fat diet for 4 weeks each. We hypothesize that patients with unexplained ADH may have an exaggerated cholesterol response to saturated fat intake. The specific aim of this study is to quantify the increase in LDL-C in unexplained ADH patients compared to FH patients. The pilot study proposed here will develop preliminary data to be used for future funding proposals of larger, randomized studies.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, age > 18 years or < 80 years
2. Pre-treatment LDL-C greater than the 95th percentile for age and sex (corresponding to 190 mg/dL for most adults), with one of the 2 following criteria: (1) tendon xanthoma (proband or first-degree relative) or (2) either first-degree relative with premature CHD (age less than 55 years in men or 65 years in women) or pretreatment LDL-C greater than the 95th percentile for age and sex.
3. Willing to come off medical therapy 4 weeks before and during study.
4. Willing to follow high/low saturated fat diet
5. Willing to attend dietary counseling sessions
6. Willing to attend frequent clinic visits
7. Subjects willing to participate under the conditions described in the informed consent form (ICF) and able to sign the ICF and applicable HIPAA forms.

Exclusion Criteria:

1. Presence of any clinically significant uncontrolled endocrine disease known to influence serum lipids or lipoproteins. Note: patients on thyroid replacement therapy can be included if the dosage of thyroxine has been stable for 6 weeks prior to the first study visit and thyroid-stimulating hormone (TSH) level is within the normal range.
2. Conditions of severe acute vascular stress (e.g. acute coronary syndrome, ischemic stroke, or major vascular surgery) within 3 months prior to the first study visit.
3. Patients unable to maintain their current activity level or planning to increase their activity level (e.g. new exercise regimen).
4. Pregnant or breast-feeding women.
5. Major illness
6. Secondary cause of dyslipidemia (e.g. obstructive liver disease, hypothyroidism, or nephrotic syndrome)
7. Hospitalization within 3 months
8. Substance abuse (illegal drug use, chronic alcoholism or problematic use of alcohol or total daily alcohol intake >2 drinks per day in men and > 1 drink per day in women).
9. Immunodeficiency or HIV-positive status
10. Illiteracy
11. Severe medical condition that may impair the ability of the person to participate in a nutrition intervention study (e.g. digestive disease with fat intolerance, advanced malignancy, or major neurological, psychiatric or endocrine disease)
12. Any other medical condition thought to limit survival to less than 1 year
13. Difficulties or major inconvenience to change dietary habits
14. History of food allergy with hypersensitivity to any of the components of olive oil or nuts

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in LDL-cholesterol | 4 weeks
  To quantify the change in low density lipoprotein cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No